CLINICAL TRIAL: NCT04276363
Title: Families, Children and Teachers Thriving Together
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-00707
Record Dates: First submitted 2019-10-02; First posted 2020-02-19 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Social Anxiety; Emotional Stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thrive Professional Learning plus ParentCorps (Experimental): 1) Professional Development, Program Training and Coaching; 2) Program for Parents of Pre-K Students; and 3) Program for Pre-K Students. The three intervention components are expected to strengthen relationships and communication between parents and teachers and promote safe, nurturing and predictable environments, which contribute to child mental health and achievement.
  Interventions: Behavioral: Thrive Professional Learning plus ParentCorps
- Thrive Professional Learning only (Experimental): Best practices in Family Engagement and Social Emotional Learning and includes an experiential approach to behavior change that asks learners to take the perspective of others and consider their own beliefs and assumptions about students, families, teachers and leaders.
  Interventions: Behavioral: Thrive Professional Learning only
- Inspire Professional Learning (Experimental): Led by the NYC Department of Education. Professional Learning sessions are tailored to the needs of pre-K teachers and leaders, and include topics aligned with the district's quality standards that support child instructional goals.
  Interventions: Behavioral: Inspire Professional Learning

INTERVENTIONS:
Behavioral: Thrive Professional Learning plus ParentCorps — led by the NYC Department of Education. Professional Learning sessions are tailored to the needs of pre-K teachers and leaders, and include topics aligned with the district's quality standards that support child instructional goals.
  Arms: Thrive Professional Learning plus ParentCorps
Behavioral: Thrive Professional Learning only — Part of the Professional Learning Track system for all Pre-K for All teachers and leaders. The NYC DOE schedules Thrive Professional Learning training days for staff on non-attendance days. Teachers attend four Professional Learning days annually, and leaders attend three days annually, over a two-year period.
  Arms: Thrive Professional Learning only
Behavioral: Inspire Professional Learning — Delivered to leaders in groups of 20 - 40 three times a year over the same two-year period. Content covers best practices in Family Engagement and Social Emotional Learning and includes an experiential approach to behavior change that asks learners to take the perspective of others and consider their own beliefs and assumptions about students, families, teachers and leaders
  Arms: Inspire Professional Learning

SUMMARY:
The current study examines the impact of ParentCorps in high-poverty district schools in New York City (NYC). The study is conducted within the context of the NYC Department of Education (DOE) Pre-K Thrive initiative. As part of this initiative, the Center for Early Childhood Health and Development (CEHD) at NYU Langone Health is implementing services to strengthen family engagement and support parents and teachers in creating safe, nurturing and predictable environments for young children. All parents of Pre-K students in the 81 district schools will be invited for them and their Pre-K children to participate in the study, which includes 2 school-based assessments in Pre-K over a 10-month period and 1 school-based assessment at the end of Kindergarten, and teacher ratings of children in Pre-K and Kindergarten. Additionally, parents will be invited to consent to the use of their children's NYC DOE administrative records from Pre-K through grade 5 for the purposes of this study. Parents will also be invited to participate by completing surveys with NYU study staff. Parents will be consented to complete two surveys when their child is in Pre-K. Parents may be randomly selected to complete a third survey when their child is in Kindergarten or to participate in a focus group with other parents.

ELIGIBILITY:
Inclusion Criteria:

* Site Selection Criteria A total of 81 of these district schools with pre-K programs in high poverty NYC neighborhoods were selected for the study in late Spring 2017 by the NYC Department of Education (DOE), following a detailed methodology developed collaboratively by the NYC DOE and NYU Investigators.

Schools must meet the following criteria:

1. have 2 or more PKFA classrooms;
2. serve a high-need population and
3. leaders ranked Thrive or Inspire as a first or second preference for the school. Sites that were currently implementing ParentCorps at the time of the randomization were not eligible for the study.

Participant Selection Criteria

* Pre-K students and families who are in the schools in 2018-2019.
* Only parents and students who are English or Spanish speaking will be eligible for participation in the study.

Exclusion Criteria:

* Families in sites other than the 81 district schools randomized to this study are excluded.
* Parents or students who do not speak English and/or Spanish will not be eligible to participate.
* Teachers and principals from the 81 sites are not considered participants in the study of student and family outcomes.

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Score on Receptive One-Word Picture Vocabulary Test (ROWPVT) | 84 Months
  A higher score indicates higher academic skills. The assessment will take 10-20 minutes - the assessor will state a word in English or Spanish, while the child is shown four images. The child must choose the image that represents the word the assessor said.
Score on Dimensional Change Card Sort (DCCS) Assessment | 84 Months
  Children are presented with a series of cards depicting images that vary along two dimensions: color and shape. Children are first asked to sort the cards by one dimension (color). After they do this for several trials, they are then asked to sort the cards by the other dimension (shape). Scores are reported as a binary "yes" or "no" - yes - child can shift to sorting by the second dimension accurately.
Score on Pencil Tap Assessment | 84 Months
  Children are asked to tap on a table twice with a pencil with the experimenter taps once, and once when the experimenter taps twice. Scores are reported as proportion of trials children answer correctly out of 16 (i.e. 1/16, 2/16, 3/16, etc.)
Score on Parental Engagement of Families Questionnaire (PEFL) | 84 Months
  The items from the PEFL questionnaire will be reported as 4-point rating scale (i.e. 1 - never, 2 - rarely, 3 - sometimes, 4 - frequently) to indicate frequency of parental engagement

SECONDARY OUTCOMES:
Score on Assessment of Children's Emotional Skills (ACES) | 84 months
  Children are presented with a series of photographs of children making happy, sad, mad, scared, or ambiguous facial expressions. For each photograph, children are asked to name the emotion expressed in the face. The higher the score indicates higher ability to match emotions.
Score on Emotion Recognition Questionnaire (ERQ) | 84 months
  16 scenarios that elicit happy, sad, mad, or scared emotions are presented to children, along with black and white line drawings to aid with comprehension (e.g. Johnny's little brother broke his toy on purpose). Children are asked to name the emotion the main character would be feeling in that situation. Scores are reported as the proportion of correct matches out of 16 (i.e. 1/16, 2/16, etc.)
Score on Patient Health Questionnaire (PHQ-9) | 84 months
  Four items are rated on a 4-point scale, ranging from 0 = not at all to 3 = nearly every day.
  This will be used to assess parent well-being.
Score on Financial Stress Questionnaire | 84 months
  To examine the degree to which parents worry about their finances, 8 questions will be asked to form a composite measure of financial stress. Parents respond to each item on a 5-point Likert scale. 5 indicates a high level of financial stress.
Score on PROMIS-10 Survey | 84 months
  10-item survey that assess general parent well-being. Participants are asked to respond on a 5-point scale, ranging from 1 (poor) to 5 (excellent)
Score on PROMIS-4 Sleep Disturbance Survey | 84 months
  This is a 4-item questionnaire assessing the quality of adult sleep. Participants are asked to respond on a 5-point scale ranging from 1 (not at all) to 5 (very much) to questions regarding their sleep quality.

OTHER OUTCOMES:
Child body mass index (BMI) | 84 months
  Children's height and weight will be measured in order to calculate BMI. The height will be measured using a stadiometer, and the weight will be measured using an electronic scale.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Brotman, MD, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to Andrea.Troxel@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.